CLINICAL TRIAL: NCT01308437
Title: An Open Label,Randomized,Comparison of the Immunogenicity and Safety of Wockhardt's Human Insulin Basal Bolus Regimen With the Novo Nordisk's Yeast Based Human Insulin Basal Bolus Regimens, Marketed in United States, in Type 1 Diabetics.
Brief Title: Immunosafety Study of Recombinant Human Insulins in Type 1 Diabetics
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Wockhardt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P3-WOS-IMS-01
Record Dates: First submitted 2011-02-09; First posted 2011-03-04 (Estimated); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Type I Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wosulin (N or 70/30 with R) (Experimental): Basal bolus conventional Insulin viz. Wosulin (N or 70/30 with R) to be injected subcutaneously.
  Interventions: Biological: Wosulin (N or 70/30 with R)
- Novolin® (N or 70/30 with R) (Active Comparator): Basal bolus conventional Insulin viz. Novolin® (N or 70/30 with R) to be injected subcutaneously.
  Interventions: Biological: Novolin® (N or 70/30 with R)

INTERVENTIONS:
Biological: Wosulin (N or 70/30 with R) — Basal bolus conventional Insulin viz. Wosulin (N or 70/30 with R) to be injected subcutaneously.
  Other Names: Wosulin R,; Wosulin N,; Wosulin 70/30
  Arms: Wosulin (N or 70/30 with R)
Biological: Novolin® (N or 70/30 with R) — Basal bolus conventional Insulin viz. Novolin® (N or 70/30 with R) to be injected subcutaneously.
  Other Names: Novolin® R,; Novolin® N,; Novolin® 70/30
  Arms: Novolin® (N or 70/30 with R)

SUMMARY:
This is an open label, randomized, parallel group comparison of the immunogenicity safety of Wockhardt's human insulin and isophane insulin compared with the Novo Nordisk's yeast based human insulin products (marketed in USA) in type 1 diabetics.

There are two phases of the study, which are as follows:

1. Phase 1 is a comparative phase in which there will be 2 arms (which are described in the section below).
2. Phase 2 is a follow up phase only applicable to Wosulin Arm.

The study will last for 54 weeks for the patients enrolled in Wosulin arm and approximately 28 weeks for the patients enrolled in the comparator arm.

Two hundred and forty two patients will be enrolled considering an estimated dropout rate of 15% for a sample size of approximately 105 evaluable patients per arm. The total planned enrollment period for this study is approximately 3 months (90 days).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who understand the nature of the study and are willing to provide written informed consent.
2. Subjects who have been pre-diagnosed as cases of type-1 diabetes (fasting C-peptide < 0.5 nmol/L) and have been on an insulin regimen for at least 12 months prior to inclusion in the trial.
3. Subjects who have been on a stable regimen of recombinant human insulin or analogs for at least 3 months prior to randomization. (A stable regimen is defined as the dose within +/- 10%).
4. Male or female subjects ≥ 18 and < 55 years of age.
5. Subjects with body mass index (BMI) of ≥18.0 to < 35.0 kg/m2
6. Subjects with glycosylated hemoglobin (HbA1c) levels between ≥6.5 and < 9.5%
7. Subjects who are cooperative, reliable, and agree to have regular injections of insulin and are willing to comply with protocol procedures.
8. Female subjects who are not pregnant and non-lactating with adequate protection from conception and fulfilling one of the following criteria are also eligible if within ≥ 18 and < 55 years age limits:

   1. Women of childbearing potential on an acceptable method of birth control (including but not limited to barrier-method, contraceptives, or intrauterine device)
   2. Women with history of bilateral tubal ligation,
   3. Women who have undergone total hysterectomy
   4. Women who are two years post-menopausal
9. Subjects who are able to use the self glucose-monitoring device and to self inject insulin.

Exclusion Criteria:

1. Female subjects who are pregnant (as confirmed by a positive urine and serum β-HCG) or are currently breast-feeding.
2. Compromised hepatic or renal function, as shown by but not limited to:

   i.Baseline AST or ALT >3 times the upper limit of normal range, and/or ii.Serum Creatinine >2.0 mg/dl and/or iii.BUN >30 mg/dl Abnormal laboratory findings will be discussed with the medical monitor prior to the subject's entry.
3. Employee of Investigator or have direct involvement with trial or other trials under the direction of Investigator.
4. Those treated with other investigational agents or devices within previous 30 days, from screening, have planned use of an investigational drug or device, or have been previously randomized in this trial.
5. History or evidence of allergy to insulin preparations.
6. History or evidence of severe hypoglycemia (severe hypoglycemic episode defined as the subject required glucose, glucagon, orange juice etc administered by a second person)
7. Requirement for total daily dose of insulin is >1.4 units/kg
8. Who have received Wockhardt's (Wosulin) or Novo Nordisk's Insulin (Novolin® R, Novolin® N, Novolin® 70/30, in US and Actrapid® Insulatard®, and Mixtard® in India) during the previous one year.
9. Serum AIA level > 20 microU/ml.
10. Receipt of any insulin of an animal origin during the last 3 years.
11. Currently receiving or have received within the last year any immunomodulators medications, including corticosteroids that would possibly modify antibody generation either at the enrollment or during the course of the study. (Topical/ ophthalmic/intra-articular/nasal spray corticosteroids will be allowed).
12. Hepatitis B or Hepatitis C or HIV positive.
13. Oral hypoglycaemic agent within 4 weeks prior to signing the consent form.
14. Who have undergone pancreatectomy or pancreas/islet cell transplant.
15. Unlikely to comply with the study protocol e.g. unable to return periodically for subsequent visits.
16. History or evidence of active severe proliferative retinopathy, nephropathy and/or neuropathy significant cardiovascular disease, anemia or hemoglobinopathy, uncontrolled hypothyroidism or uncontrolled hyperthyroidism, alcohol or drug abuse or any other medical condition that in the opinion of Investigator can interfere with the study.
17. Judged by the investigator as inappropriate to participate in the study for any reason other than those mentioned above.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 134 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in HbAlc from baseline to 6 months of treatment between Wosulin arm and Novolin arm(as surrogate indicator of change in insulin antibodies titers between the two treatment arms). | 6 months

SECONDARY OUTCOMES:
Correlation between change in HbA1c and change in anti insulin and insulin neutralizing antibodies. | 6 months and 12 months
  Insulin dose will be used as a covariate
To compare the change from baseline in the level of serum anti insulin antibodies and insulin neutralizing antibodies between the two arms | 6 months
Compare the change in Insulin dose between the two arms | 3 and 6 months
  Glycated hemoglobin levels and the number of hypoglycemic episodes will be the covariants for this analysis
Correlation of the immunogenicity with hypoglycemia, local allergic reactions and systemic allergic reactions will be evaluated. | 6 and 12 months
  Immunogenicity is measured as percentage change in serum antiinsulin antibodies and insulin neutralizing antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Ashima Bhatia, M.D., Study Director — Wockhardt
Locations (25):
- United States (17):
  - University Clinical Investigators, Inc. dba Diabetes Research Center, Tustin, California
  - International Research Associates, Hialeah, Florida
  - The Center for Diabetes and Endocrine Care, Hollywood, Florida
  - Baptist Diabetes Associates, PA, Miami, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Ormond Medical Arts Pharmaceutical Research Center, Ormond Beach, Florida
  - Suncoast Clinical Research, Palm Harbor, Florida
  - International Clinical Research - US, LLC, Sanford, Florida
  - Cotton-O'Neil Clinical Research Center, Diabetes & Endocrinology, Topeka, Kansas
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - Endocrine & Metabolic Consultants, Rockville, Maryland
  - ActivMed Practices and Research, Haverhill, Massachusetts
  - Alzohaili Medical Consultants, Dearborn, Michigan
  - ActivMed Practices and Research, Rochester, New Hampshire
  - University Diabetes & Endocrine Association, Chattanooga, Tennessee
  - Sergio Rovner, MD, El Paso, Texas
  - Optimum Clinical Research, Inc., Salt Lake City, Utah
- India (8):
  - Dr Rakesh Sahay, Hyderabad, Andhra Pradesh
  - Dia Care - A Complete Diabetes Care Centre, Ahmedabad, Gujarat
  - Dr Sanjay Kalra, Karnāl, Haryana
  - Dr Mala Dharmalingam, Bangalore, Karnataka
  - Bangalore Diabetes Hospital, Bangalore, Karnataka
  - Dr Sharad Pendsey, Nagpur, Maharashtra
  - Diabetes Thyroid &Endocrine Centre, Jaipur, Rajasthan
  - Bhandari's Clinic, Jaipur, Rajasthan